CLINICAL TRIAL: NCT07248618
Title: Comparison of Trunk Training Exercises and Lateral Truncal Tilt Balance Training on Trunk Control, Balance and Activities of Daily Living in Stroke Patients
Brief Title: Comparison of TTE and LTTBT on Trunk Control, Balance and ADL's in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/02102
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trunk Training Exercises (Active Comparator): Core Stabilization Exercises, dynamic trunk exercises, bridging exercises
  Interventions: Other: Trunk Training Exercises
- Lateral Truncal Tilt Balance Training (Experimental): Seated lateral tilts, Standing Lateral Weight Shifts, balance board tilts, Stability Ball Exercises, lateral Reaches on Unstable Surface
  Interventions: Other: Lateral Truncal Tilt Balance Training

INTERVENTIONS:
Other: Trunk Training Exercises — Group A will undergo a structured trunk training exercise program focused on strengthening the core muscles involved in trunk control. This program will include both dynamic and static exercises targeting trunk flexion, extension, and rotation, which are critical for improving postural stability and overall trunk coordination.
  Frequency: Sessions will be conducted three times per week for the duration of 8 weeks.
  Session Duration: Each session will last approximately 45 minutes, including a warm-up, main exercises, and a cool-down period.
  Arms: Trunk Training Exercises
Other: Lateral Truncal Tilt Balance Training — Group B will follow a lateral truncal tilt balance training program focusing on balance improvement through lateral stability exercises. This training emphasizes body tilts and weight shifts to encourage trunk control and postural alignment, particularly targeting the common lateral asymmetries observed in stroke patients.
  Frequency: Sessions will be conducted three times per week for 8 weeks. Session Duration: Each session will last approximately 45 minutes, including warm-up, main exercises, and a cool-down period.
  Arms: Lateral Truncal Tilt Balance Training

SUMMARY:
To compare the effects of trunk training exercises and lateral truncal tilt balance training on trunk control, balance and activities of daily living in stroke patients.The primary outcome measures used to evaluate the efficacy of each training approach will include the Timed Up and Go (TUG) test, assessing mobility and fall risk; the Berg Balance Scale (BBS), which measures functional balance; and the Trunk Impairment Scale (TIS), evaluating trunk control and coordination.

DETAILED DESCRIPTION:
Stroke is a significant cause of disability globally, affecting millions each year. Stroke patients frequently experience impairments in trunk control and balance, critical factors for independence in activities of daily living (ADLs). Two promising therapeutic approaches include Trunk Training Exercises (TTE) focusing on core stability and Lateral Truncal Tilt Balance Training (LTT), which targets balance and postural alignment through controlled lateral movements. This study aims to compare the effectiveness of these two interventions in improving trunk control, balance, and ADLs in stroke patients, potentially leading to optimized rehabilitation practices. A randomized clinical trial will be conducted at Jinnah Hospital, Lahore. Participants aged 40 75, diagnosed with sub-acute stroke, will be randomly assigned to one of two groups: Group A, which will undergo trunk training exercises (TTE), and Group B, which will receive lateral truncal tilt balance training (LTT). Each intervention will last for eight weeks and thrice a week, with a session of 45 minutes including warm-up exercises, main exercises and cool down period during which participants will engage in their respective training regimens. To assess the impact of these interventions, baseline measurements will be taken prior to the intervention and compared to post-intervention results. The primary outcome measures used to evaluate the efficacy of each training approach will include the Timed Up and Go (TUG) test, assessing mobility and fall risk; the Berg Balance Scale (BBS), which measures functional balance; and the Trunk Impairment Scale (TIS), evaluating trunk control and coordination. Data analysis will be conducted using SPSS software (version 25). To determine the distribution of data, the Shapiro-Wilk Test will be performed. If the data is not normally distributed, the Wilcoxon Signed Rank Test will be used to analyze within-group differences, while the Mann-Whitney U Test will assess differences between groups at each interval. For normally distributed data, Paired Sample T-tests will compare pre- and post-intervention scores within each group, and Independent Sample T-tests will evaluate changes between groups.

Inclusion criteria is:

Patients with ischemic stroke Both male and females Age 40-75 years Patients diagnosed with sub-acute stroke after six months to 1.5 years of diagnosis Patients able to walk 10 meters independently Score less than 21 on trunk impairment scale Patients with score 24 or more on MMSE

Exclusion criteria is:

Patients with score more than 2 on modified Ashworth scale will be excluded Chronic patients will not be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic stroke
* Both male and females
* Age 40-75 years
* Patients diagnosed with sub-acute stroke after six months to 1.5 years of diagnosis
* Patients able to walk 10 meters independently
* Score less than 21 on trunk impairment scale
* Patients with score 24 or more on MMSE

Exclusion Criteria:

* Patients with score more than 2 on modified Ashworth scale will be excluded
* Chronic patients will not be included in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Timed up and go test (TUG) | 1-2 min
  The Timed Up and Go (TUG) test is a simple and widely used assessment to evaluate a person's mobility, balance, and risk of falling, particularly in older adults and individuals with neurological conditions like stroke. A time of under 10 seconds is typically considered normal for healthy adults, while times over 12-14 seconds may indicate a higher risk of falls and impaired mobility. It has good validity and reliability ranging from 0.80-0.83

SECONDARY OUTCOMES:
Berg balance scale (BBS) | 15 to 20 min
  . The scale consists of 14 functional tasks, such as standing from a seated position, reaching forward, standing with eyes closed, and turning 360 degrees. Each task is scored on a 5-point scale from 0 (unable to perform) to 4 (normal performance), yielding a maximum score of 56, with lower scores indicating a greater risk of falling (20).

OTHER OUTCOMES:
Trunk impairment scale (TIS) | upto 20 min
  . It includes three subscales: static sitting balance, dynamic sitting balance, and trunk coordination, with scores ranging from 0 to 23 points, where higher scores indicate better trunk stability and coordination

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Jinnah hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tu WJ, Wang LD; Special Writing Group of China Stroke Surveillance Report. China stroke surveillance report 2021. Mil Med Res. 2023 Jul 19;10(1):33. doi: 10.1186/s40779-023-00463-x. PMID 37468952
- [Background] Murphy SJ, Werring DJ. Stroke: causes and clinical features. Medicine (Abingdon). 2020 Sep;48(9):561-566. doi: 10.1016/j.mpmed.2020.06.002. Epub 2020 Aug 6. PMID 32837228
- [Background] Lee K. The Relationship of Trunk Muscle Activation and Core Stability: A Biomechanical Analysis of Pilates-Based Stabilization Exercise. Int J Environ Res Public Health. 2021 Dec 4;18(23):12804. doi: 10.3390/ijerph182312804. PMID 34886530
- [Background] Karthikbabu S, Verheyden G. Relationship between trunk control, core muscle strength and balance confidence in community-dwelling patients with chronic stroke. Top Stroke Rehabil. 2021 Mar;28(2):88-95. doi: 10.1080/10749357.2020.1783896. Epub 2020 Jun 23. PMID 32574524
- [Background] Pellicciari L, Sodero A, Campagnini S, Guolo E, Basagni B, Castagnoli C, Hochleitner I, Paperini A, Gnetti B, Avila L, Romano E, Grippo A, Hakiki B, Carrozza MC, Mannini A, Macchi C, Cecchi F. Factors influencing trunk control recovery after intensive rehabilitation in post-stroke patients: a multicentre prospective study. Top Stroke Rehabil. 2023 Mar;30(2):109-118. doi: 10.1080/10749357.2021.2016099. Epub 2022 Jan 7. PMID 34994302
- [Background] Martins LG, Molle da Costa RD, Alvarez Sartor LC, Thomaz de Souza J, Winckler FC, Regina da Silva T, Modolo GP, Nunes HRC, Bazan SGZ, Martin LC, Luvizutto GJ, Bazan R. Clinical factors associated with trunk control after stroke: A prospective study. Top Stroke Rehabil. 2021 Apr;28(3):181-189. doi: 10.1080/10749357.2020.1805244. Epub 2020 Aug 10. PMID 32772828
- [Background] Lee K, Lee D, Hong S, Shin D, Jeong S, Shin H, Choi W, An S, Lee G. The relationship between sitting balance, trunk control and mobility with predictive for current mobility level in survivors of sub-acute stroke. PLoS One. 2021 Aug 5;16(8):e0251977. doi: 10.1371/journal.pone.0251977. eCollection 2021. PMID 34351943
- [Background] Sawa K, Amimoto K, Ishigami K, Miyamoto T, Setoyama C, Suzuki R, Nozomi K, Tamura M, Miyagami M. Efficacy of lateral truncal tilt training with a wedge on postural vertical and activities of daily living in recovery phase after stroke: A randomized crossover trial. NeuroRehabilitation. 2022;51(1):33-40. doi: 10.3233/NRE-210255. PMID 35275567
- [Background] De Luca A, Squeri V, Barone LM, Vernetti Mansin H, Ricci S, Pisu I, Cassiano C, Capra C, Lentino C, De Michieli L, Sanfilippo CA, Saglia JA, Checchia GA. Dynamic Stability and Trunk Control Improvements Following Robotic Balance and Core Stability Training in Chronic Stroke Survivors: A Pilot Study. Front Neurol. 2020 Jun 17;11:494. doi: 10.3389/fneur.2020.00494. eCollection 2020. PMID 32625162
- [Background] Shalash A, Fayed ZY, Hamid E, Radwan H, Nada MA, Eid M, Abdel Ghany WA. Outcome of pallidal stimulation of idiopathic generalized dystonia with predominant mobile truncal dystonia: case report. Int J Neurosci. 2022 May;132(5):429-433. doi: 10.1080/00207454.2020.1818743. Epub 2020 Sep 16. PMID 32886009
- [Background] Tamura S, Miyata K, Kobayashi S, Takeda R, Iwamoto H. The minimal clinically important difference in Berg Balance Scale scores among patients with early subacute stroke: a multicenter, retrospective, observational study. Top Stroke Rehabil. 2022 Sep;29(6):423-429. doi: 10.1080/10749357.2021.1943800. Epub 2021 Jun 25. PMID 34169808
- [Background] Jin X, Wang L, Liu S, Zhu L, Loprinzi PD, Fan X. The Impact of Mind-body Exercises on Motor Function, Depressive Symptoms, and Quality of Life in Parkinson's Disease: A Systematic Review and Meta-analysis. Int J Environ Res Public Health. 2019 Dec 18;17(1):31. doi: 10.3390/ijerph17010031. PMID 31861456